CLINICAL TRIAL: NCT00394212
Title: Randomized Evaluation of Endoscopic Suturing Transorally for Anastomotic Outlet Reduction (RESTORe) for Patients With Inadequate Weight Loss Following Roux-en-Y Gastric Bypass Surgery
Brief Title: Incisionless Treatment for Patients With Inadequate Weight Loss Following Roux-en-Y Gastric Bypass
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: For business reasons
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DVL-EC-002
Record Dates: First submitted 2006-10-27; First posted 2006-10-31 (Estimated); Results first posted 2012-11-07 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2012-10

CONDITIONS: Obesity
Keywords: Weight Loss; Transoral Suturing; Dilated gastrojejunostomy; Inadequate weight loss following primary RYGB
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Transoral suturing of the dilated gastrojejunostomy
  Interventions: Device: Transoral Suturing
- 2 (Sham Comparator): Sham Endoscopy (suturing not performed)
  Interventions: Other: Sham Endoscopy

INTERVENTIONS:
Device: Transoral Suturing — suturing of anastomosis
  Arms: 1
Other: Sham Endoscopy — suturing not performed
  Arms: 2

SUMMARY:
It is estimated that up to 20% of patients who have Roux-en-Y Gastric Bypass (RYGB) surgery will not meet their weight loss goal, or may even regain some of the weight they initially lost. One possible explanation is that the opening between the stomach pouch and the intestine becomes stretched. If this opening becomes too wide, food may be able to pass from the stomach to the intestine too quickly - causing patients to feel less full after eating.

For some patients, doctors may recommend additional invasive surgery to tighten the opening between the stomach pouch and the small intestine. Although this may help patients resume their weight loss, the risk of complications during a second surgical procedure is significantly higher than the risk during the original gastric bypass.

The purpose of this study is to evaluate an incisionless procedure for patients who have either had inadequate weight loss or have regained weight following gastric bypass. The procedure is designed to tighten the opening between the stomach pouch and the small intestine, which may slow down the passage of food to help patients feel full longer after eating.

ELIGIBILITY:
Inclusion Criteria:

* 6 months post primary RYGB with inadequate weight loss or weight regain
* BMI >30 and ≤ 50
* Dilated gastrojejunal anastomosis
* Successfully completes screening process
* Signed consent

Exclusion Criteria:

* Recently quit smoking or plan to quit within the next year
* Pregnant or planning to become pregnant over the course of the next 9 months
* Mallampati score of 4
* Serious systemic disease or active disease of the gastrointestinal tract
* Gastric pouch abnormalities
* Significant movement limitations
* Use of weight-promoting or weight-reduction drugs during study period
* Severe eating disorders
* Uncontrolled depression or psychoses
* Ongoing severe complication resulting from initial RYGB or other condition that in the investigators' assessment would make the patient an unsuitable candidate for the study procedure
* History of significant cardiovascular, cerebrovascular or pulmonary disease
* Not a candidate for conscious or general sedation
* Anticoagulant therapies
* Active substance abuse
* Life expectancy < 1 year
* Enrolled in another investigational drug or device trial that has not completed the primary endpoint or that clinically interferes with this trial's study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2006-11; Primary Completion 2008-09 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Denver, Colorado
  - Baltimore, Maryland
  - Boston, Massachusetts
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - New York, New York
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Thompson CC, Chand B, Chen YK, DeMarco DC, Miller L, Schweitzer M, Rothstein RI, Lautz DB, Slattery J, Ryan MB, Brethauer S, Schauer P, Mitchell MC, Starpoli A, Haber GB, Catalano MF, Edmundowicz S, Fagnant AM, Kaplan LM, Roslin MS. Endoscopic suturing for transoral outlet reduction increases weight loss after Roux-en-Y gastric bypass surgery. Gastroenterology. 2013 Jul;145(1):129-137.e3. doi: 10.1053/j.gastro.2013.04.002. Epub 2013 Apr 5. PMID 23567348

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at bariatric centers of excellence with screening initiated on 25Oct2006. The first randomized procedure was performed on 3Apr2007. The last subject follow-up was performed 8May2009.
Pre-assignment Details: Prior to enrollment, prospective candidates having provided informed consent were screened for eligibility during a formal 6 week screening period. Screening performed by a multidisciplinary team including surgeon and/or endoscopist, psychiatric professional and registered dietician.
Groups:
- EndoCinch Suturing System:Transoral Suturing: Transoral suturing of the dilated gastrojejunostomy
- Sham Endoscopy: Sham Endoscopy (suturing not performed)
Period: Overall Study
Arm/Group | EndoCinch Suturing System:Transoral Suturing | Sham Endoscopy
Started | 50 (2 subjects assigned to suturing underwent sham procedure, results based on Intent-To-Treat (ITT)) | 27
6 Week Follow-up | 45 | 26
3 Month Follow-up | 45 | 26
6 Month Follow-up | 43 | 26
Completed | 43 | 26
Not Completed | 7 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EndoCinch Suturing System:Transoral Suturing | Sham Endoscopy | Total
Number analyzed (Participants) | 50 | 27 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 27 | 76
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (9.5) | 47.6 (7.0) | 47.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 26 | 73
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 50 | 27 | 77

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss (%)
Description: Percent Weight Loss is computed as [(Baseline weight - 6 mo. weight) / Baseline weight] * 100
Time Frame: 6 months
Population: ITT using Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: percentage of weight lost
Arm/Group | EndoCinch Suturing System:Transoral Suturing | Sham Endoscopy
Number analyzed (Participants) | 50 | 27
percentage of weight lost | 4.2 (5.4) | 1.9 (5.2)
Statistical Analysis 1: Comparison: EndoCinch Suturing System:Transoral Suturing vs Sham Endoscopy; Based on a 2-group test of means for unequal variance and unequal sample size (2:1 randomization ratio) with alpha = 0.05 and a power of 80%, the sample size required was 132; 88 subjects in the Transoral Suturing arm and 44 in the Sham Endoscopy arm. The study was prematurely discontinued due to reasons unrelated to safety and effectiveness and therefore was underpowered for evaluation of the primary and secondary hypotheses; Test type: Superiority or Other; p = 0.066, Wilcoxon (Mann-Whitney) — P-value from non-parametric Mann-Whitney-Wilcoxon test comparing treatments

2. Secondary Outcome: Subjects Achieving 15% Excess Weight Loss (EWL)
Description: %Excess Weight Loss (%EWL) is computed as:[(Weight at Baseline - Weight at 6 months)/(Weight at Baseline - Ideal Weight at BMI of 25)]*100.
Time Frame: 6 months
Population: ITT, Last Observation Carried Forward
Measure: Number; unit: percentage of participants
Arm/Group | EndoCinch Suturing System:Transoral Suturing | Sham Endoscopy
Number analyzed (Participants) | 50 | 27
percentage of participants | 41.3 | 25.9
Statistical Analysis 1: Comparison: EndoCinch Suturing System:Transoral Suturing vs Sham Endoscopy; Test type: Superiority or Other; p = 0.317, Fisher Exact — P-value from two-sided Fisher's exact test comparing percents achieving 15% EWL at 6 months for the two treatments

3. Secondary Outcome: Subjects Achieving Weight Stabilization at 6 Months
Description: Weight is stabilized if 6 month weight is +/- 2% from baseline weight.
Time Frame: 6 months
Population: ITT, Last Observation Carried Forward
Measure: Number; unit: percentage of participants
Arm/Group | EndoCinch Suturing System:Transoral Suturing | Sham Endoscopy
Number analyzed (Participants) | 50 | 27
percentage of participants | 96.0 | 77.8
Statistical Analysis 1: Comparison: EndoCinch Suturing System:Transoral Suturing vs Sham Endoscopy; Test type: Superiority or Other; p = 0.019, Fisher Exact — P-value from two-sided Fisher's exact test comparing percents achieved for the two treatments

4. Secondary Outcome: Subjects Achieving 20% Excess Weight Loss at 6 Months
Description: %Excess Weight Loss (%EWL) is computed as: [(Weight at Baseline - Weight at 6 months)/(Weight at Baseline - Ideal Weight at BMI of 25)]*100
Time Frame: 6 months
Population: ITT, Last Observation Carried Forward
Measure: Number; unit: percentage of participants
Arm/Group | EndoCinch Suturing System:Transoral Suturing | Sham Endoscopy
Number analyzed (Participants) | 50 | 27
percentage of participants | 33.3 | 14.8
Statistical Analysis 1: Comparison: EndoCinch Suturing System:Transoral Suturing vs Sham Endoscopy; Test type: Superiority or Other; p = 0.174, Fisher Exact — P-value from two-sided Fisher's exact test comparing percents achieved for the two treatments

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | EndoCinch Suturing System:Transoral Suturing | Sham Endoscopy
Serious Adverse Events (participants affected / at risk) | 2/48 | 0/29
Other Adverse Events (participants affected / at risk) | 18/48 | 10/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoCinch Suturing System:Transoral Suturing (N=48) | Sham Endoscopy (N=29)
Adhesion-related intestinal obstruction (from prior surgery) (Gastrointestinal disorders) | 1 (1) | 0 (0) — Adhesion from initial gastric bypass surgery
Pulmonary edema secondary to fluid overload (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — edema secondary to fluid overload following study procedure
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoCinch Suturing System:Transoral Suturing (N=48) | Sham Endoscopy (N=29)
Nausea (Gastrointestinal disorders) | 8 (9) | 3 (3)
Vomiting (Gastrointestinal disorders) | 6 (6) | 4 (5)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4)
Abdominal Discomfort (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Headache (Nervous system disorders) | 3 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of this study are that study enrollment was prematurely discontinued; therefore the study was underpowered for the analysis of both the primary and secondary effectiveness endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
First publication of study results will be the multicenter results. In the event no multicenter publication has been made within one to two years of the completion of the study at all centers, Investigators will be free to publish their own single-center results. Investigators seeking publication must submit a draft for sponsor review at least 60 days prior to submission of the draft for publication. Sponsor cannot require changes to the communication and cannot extend the embargo.